CLINICAL TRIAL: NCT00292279
Title: The Impact of Omega-3 Fat Emulsion on Clinical Outcome of Post-Operative Cancer Patients: A Randomized, Double Blind, Controlled, Multi-Center Clinical Trial.
Brief Title: The Impact of Omega-3 Fat Emulsion on Clinical Outcome of Post-Operative Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sino-Swed Pharmaceutical Corporation (Industry)
Responsible Party: TF Ye, Ethic Committee of Peking Union Medical College Hospital
Organization: Fresenius Kabi Sino-Swed Pharmaceutical Corp. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HL20020004
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Carcinoma Surgery; Parenteral Nutrition; Post-Operative Hospital Stay
Keywords: Impact of Omega 3 fatty acid on outcome; Omega-3 fatty acid; Carcinoma surgery; Digestive System; Parenteral Nutrition; Fat Emulsions, Intravenous; Clinical outcome; SIRS; Infectious complication; Postoperative hospital stay; Cost of postoperative period; Post-operative nutritional cost & total treatment cost
MeSH Terms: conditions — Hyperphagia | interventions — fish oil triglycerides; soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Omega-3 fish oil emulsion (Omegaven )
- B (Active Comparator)
  Interventions: Drug: long-chain triglyceride

INTERVENTIONS:
Drug: Omega-3 fish oil emulsion (Omegaven ) — Patients of the treatment group received 0.2 g fish oil (10% Omegaven, Fresenius Kabi, Bad Homburg, Germany) and 1.0 g soy bean oil per kg BW per day
  Other Names: Omegaven
  Arms: A
Drug: long-chain triglyceride — the control group received 1.2 g soy bean oil (Intralipid, Sino-Swed,Wuxi,China)
  Other Names: Intralipid
  Arms: B

SUMMARY:
The purpose of this study is to evaluate clinical safety and effect of Omega-3 fat oil emulsion on outcome in post-operative cancer patients.

DETAILED DESCRIPTION:
As an essential component of parenteral nutrition, fat emulsion has been used more than 30 years. It provides energy and essential fatty acids. Commercial fatty emulsion products mostly come from soy bean. The omega 6 fatty acids make up with the major fatty acids of this fat emulsion, and lack of omega 3 fatty acids generally. The imbalance of these two types of fatty acids may impact with negative clinical outcomes.

There are lots of omega 3 fatty acids makes up with fish oil emulsion, especially with eicosapentaenoic acid (EPA) and Docosahexaenoic acid (DHA).Few clinical studies found its clinical efficacy in recently years. A commercial product of omega 3 fat emulsion by Fresenius-Kabi was registered in Europe at 1998. There is no any clinical trial in Asia to elaborate the efficacy of omega 3 fat emulsion, as well the lack of large scale clinical trial in the world.

Currently study is the first large scale, randomized, double blind and multi-center clinical trial to elaborate the impact of fish oil fat emulsion in Asia and Europe.

ELIGIBILITY:
Inclusion Criteria:

* Post-operative male and female cancer patients
* Require post operative parenteral nutrition support at least 7 days based on nutritional risk screening(BMI 20-25)
* Sign an informed consent

Exclusion Criteria:

* Diabetes Mellitus
* Abnormal fatty metabolism (TG>200mg/dl or cholesterol>240mg/dl )
* Renal dysfunction (Cr>1.6mg/dl or BUN>30mg/dl)
* Liver dysfunction (ALT>60U/L or TBIL>1.2mg/dl)
* Lienectomy
* Temperature>37.5°C
* Undergoing hormone therapy
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2002-06; Primary Completion 2003-11 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Infectious complication | POD+1 to POD+14
Systemic inflammatory response syndrome (SIRS) | POD+1 to POD +8

SECONDARY OUTCOMES:
Post-operative hospitalization days | POD+1 to discharge
Post operative nutritional cost & total treatment cost | POD+1 to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Zhu-ming Jiang, FACS, Study Director — Peking Union Medical College Hospital
Locations (5):
- China (5):
  - People's Hospital, Beijing University, Beijing
  - Beijing Friendship Hospital, Beijing
  - Beijing Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - General Hospital Of PLA, Beijing

REFERENCES:
- [Result] (Abstract) ZM Jiang, XR Wang, JM Wei, Y. Wang, Y. Li, S Wang, DW Wilmore. The impact of i.v. fish oil emulsion on clinical outcome & immune functions of post-operative cancer patients: a randomized, double blind, controlled, multi-center clinical trial for 203 cases Clinical Nutrition(Abstract for ESPEN 2005)(Absract No. 181)
- [Derived] Jiang ZM, Wilmore DW, Wang XR, Wei JM, Zhang ZT, Gu ZY, Wang S, Han SM, Jiang H, Yu K. Randomized clinical trial of intravenous soybean oil alone versus soybean oil plus fish oil emulsion after gastrointestinal cancer surgery. Br J Surg. 2010 Jun;97(6):804-9. doi: 10.1002/bjs.6999. PMID 20473991